CLINICAL TRIAL: NCT03277248
Title: Phase III: UbLiTuximab in Multiple Sclerosis Treatment Effects (ULTIMATE II STUDY)
Brief Title: Study to Assess the Efficacy and Safety of Ublituximab in Participants With Relapsing Forms of Multiple Sclerosis (RMS)
Acronym: ULTIMATE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG1101-RMS302; 2017-000639-15 (EudraCT Number)
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Relapsing Multiple Sclerosis (RMS)
MeSH Terms: interventions — ublituximab; teriflunomide

STUDY DESIGN:
Intervention Model Description: Randomized, multi-center, double-blinded, active-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded, active-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ublituximab + Oral Placebo (Experimental): Participants received ublituximab intravenous (IV) infusion, 150 milligrams (mg) over 4 hours (h) on Day 1 followed by 450 mg over 1 h on Days 15, 168, 336 and 504 (Week 72) along with the oral placebo tablet, once daily (QD) from Day 1 up to the last day of Week 95.
  Interventions: Biological: Ublituximab; Drug: Oral Placebo
- Teriflunomide + IV Placebo (Active Comparator): Participants received teriflunomide 14 mg tablet, orally, QD from Day 1 up to the last day of Week 95 along with the placebo IV infusion on Days 1, 15, 168, 336 and 504 (Week 72).
  Interventions: Drug: Teriflunomide; Drug: IV Placebo

INTERVENTIONS:
Biological: Ublituximab — Administered as an IV infusion.
  Other Names: TG-1101
  Arms: Ublituximab + Oral Placebo
Drug: Teriflunomide — Film coated tablets administered orally.
  Arms: Teriflunomide + IV Placebo
Drug: Oral Placebo — Administered orally.
  Arms: Ublituximab + Oral Placebo
Drug: IV Placebo — Administered as an IV Infusion.
  Arms: Teriflunomide + IV Placebo

SUMMARY:
This study determines the Annualized Relapse Rate (ARR) in participants with RMS after 96 weeks (approximately 2 years) treatment with intravenous (IV) infusion of ublituximab/oral placebo compared to 14 mg oral teriflunomide/IV placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing multiple sclerosis (RMS) (McDonald Criteria 2010)
* Active disease
* Expanded disability status scale (EDSS) 0 - 5.5 (inclusive) at screening

Exclusion Criteria:

* Treatment with prior Anti-cluster of differentiate 20 (CD20) or other B cell directed treatment
* Treatment with the following therapies at any time prior to randomization: alemtuzumab, natalizumab, teriflunomide, leflunomide and Stem cell transplantation
* Diagnosed with primary progressive multiple sclerosis (PPMS)
* Pregnant or nursing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 545 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - TG Therapeutics RMS Investigational Trial site, Phoenix, Arizona
  - TG Therapeutics RMS Investigational Trial Site, Aurora, Colorado
  - TG Therapeutics RMS Investigational Trial Site, Tampa, Florida
  - TG Therapeutics RMS Investigational Trial Site, Lexington, Kentucky
  - TG Therapeutics RMS Investigational Trial Site, Chesterfield, Missouri
  - TG Therapeutics RMS Investigational Trial Site, Las Vegas, Nevada
  - TG Therapeutics RMS Investigational Trial Site, Teaneck, New Jersey
  - TG Therapeutics RMS Investigational Trial Site, Albuquerque, New Mexico
  - TG Therapeutics RMS Investigational Trial Site, Patchogue, New York
  - TG Therapeutics RMS Investigational Trial site, Columbus, Ohio
  - TG Therapeutics RMS Investigational Trial Site, Pittsburgh, Pennsylvania
  - TG Therapeutics RMS Investigational Trial site, San Antonio, Texas
  - TG Therapeutics RMS Investigational Trial site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after study completion via publication.

REFERENCES:
- [Derived] Alvarez E, Steinman L, Fox EJ, Hartung HP, Qian P, Wray S, Robertson D, Selmaj K, Wynn D, Mok K, Xu Y, Bodhinathan K, Miskin HP, Cree BAC. Improvements in no evidence of disease activity with ublituximab vs. teriflunomide in the ULTIMATE phase 3 studies in relapsing multiple sclerosis. Front Neurol. 2024 Oct 24;15:1473284. doi: 10.3389/fneur.2024.1473284. eCollection 2024. PMID 39512280
- [Derived] Steinman L, Fox E, Hartung HP, Alvarez E, Qian P, Wray S, Robertson D, Huang D, Selmaj K, Wynn D, Cutter G, Mok K, Hsu Y, Xu Y, Weiss MS, Bosco JA, Power SA, Lee L, Miskin HP, Cree BAC; ULTIMATE I and ULTIMATE II Investigators. Ublituximab versus Teriflunomide in Relapsing Multiple Sclerosis. N Engl J Med. 2022 Aug 25;387(8):704-714. doi: 10.1056/NEJMoa2201904. PMID 36001711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 545 participants were enrolled across investigative sites in Belarus, Spain, the United Kingdom, Croatia, Poland, Russia, Ukraine, and the United States from 25 August 2017 to 12 November 2020.
Pre-assignment Details: A total of 629 participants were screened and of those, 545 were enrolled and randomized to receive either ublituximab/oral placebo or teriflunomide/IV placebo.
Period: Overall Study
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Started | 272 | 273
Completed (Completed = Number of participants who completed the 96 weeks Treatment Period) | 254 | 239
Not Completed | 18 | 34
Not completed — Adverse Event | 3 | 1
Not completed — Subject Withdrawal of Consent | 6 | 23
Not completed — Investigator/Sponsor Decision | 2 | 2
Not completed — Pregnancy | 4 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Other-Alternative Treatment//COVID-19 related/Unspecified Reasons | 3 | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population consisted of all randomized participants.
Groups:
- Ublituximab + Oral Placebo: Participants received ublituximab IV infusion, 150 mg over 4 h on Day 1 followed by 450 mg over 1 h on Days 15, 168, 336 and 504 (Week 72) along with the oral placebo tablet, QD from Day 1 up to the last day of Week 95.
- Total: Total of all reporting groups
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo | Total
Number analyzed (Participants) | 272 | 273 | 545
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (8.76) | 36.2 (8.97) | 35.3 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 176 | 354
  Male | 94 | 97 | 191
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 3 | 5
  White | 269 | 269 | 538
  Other | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 262 | 263 | 525
  Not Reported | 2 | 2 | 4
  Unknown | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  Belarus | 29 | 35 | 64
  Spain | 6 | 2 | 8
  United Kingdom | 4 | 1 | 5
  Croatia | 25 | 24 | 49
  Poland | 39 | 38 | 77
  Russia | 78 | 85 | 163
  Ukraine | 74 | 69 | 143
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR)
Description: ARR is defined as the number of Independent Relapse Adjudication Committee (IRAP)-confirmed relapses per participant year. The estimate of ARR for a treatment group is the total number of relapses for participants in the respective treatment group divided by the sum of treatment duration for participants in that specific treatment group.
Time Frame: Up to 96 weeks
Population: Modified Intention-to-Treat (mITT) population consisted of all participants in the ITT population who received at least one dose of study medication and had at least one baseline and post baseline efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: relapses per participant-years
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 272 | 272
relapses per participant-years | 0.091 [0.049 to 0.169] | 0.178 [0.109 to 0.291]
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p = 0.0022, Negative Binomial Model — GEE (Generalized Estimating Equation) model for the relapse count per participant with logarithmic link function, treatment, region, and baseline Expanded Disability Status Scale (EDSS) strata as covariates and log (years of treatment) as offset; Rate Ratio (Ublituximab / Teriflunomide) = 0.509, 95% CI 2-sided [0.330 to 0.784]

2. Secondary Outcome: Total Number of Gadolinium (Gd)-Enhancing T1-Lesions Per Magnetic Resonance Imaging (MRI) Scan Per Participant
Description: The total number of Gd-enhancing T1-lesions were calculated as the sum of the individual number of lesions at Weeks 12, 24, 48, and 96, divided by the total number of MRI scans of the brain.
Time Frame: Weeks 12, 24, 48, and 96
Population: mITT-MRI population consisted of participants in the mITT population who had a baseline and at least 1 post-baseline MRI efficacy assessments.
Measure: Least Squares Mean (95% Confidence Interval); unit: lesions per scan per participant
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 272 | 267
lesions per scan per participant | 0.009 [0.004 to 0.017] | 0.250 [0.162 to 0.385]
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p < .0001, Negative Binomial Model — GEE model for the relapse count per participant with logarithmic link function, treatment, region, and baseline EDSS strata as covariates and log (years of treatment) as offset; Rate Ratio (Ublituximab / Teriflunomide) = 0.035, 95% CI 2-sided [0.019 to 0.064]

3. Secondary Outcome: Total Number of New and Enlarging T2 Hyperintense Lesions (NELs) Per MRI Scan Per Participant
Description: The total number of NELs were calculated as the sum of the individual number of lesions at Weeks 24, 48, and 96, divided by the total number of MRI scans of the brain.
Time Frame: Weeks 24, 48, and 96
Population: mITT-MRI population consisted of participants in the mITT population who had a baseline and at least 1 post-baseline MRI efficacy assessments. Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: lesions per scan per participant
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 269 | 259
lesions per scan per participant | 0.282 [0.200 to 0.397] | 2.831 [2.128 to 3.767]
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p < .0001, Negative Binomial Model — [p-value comment as in outcome 2, analysis 1]; Rate Ratio (Ublituximab / Teriflunomide) = 0.100, 95% CI 2-sided [0.073 to 0.136]

4. Secondary Outcome: Time to Confirmed Disability Progression (CDP) for at Least 12 Weeks
Description: 12-week CDP is defined as an increase in EDSS at least 1 point higher than the baseline EDSS if the baseline EDSS is ≤5.5 or at least 0.5 higher than the baseline EDSS if the baseline EDSS is >5.5. The EDSS is based on a standard neurological examination, (pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, and cerebral) and ambulation function system assessments. The EDSS disability scale ranges in 0.5-point steps from 0 (normal) to 10 (death) where higher scores indicate disability. The time to onset of 12-week CDP is the time to progression to the EDSS change defined above.
Time Frame: Up to Week 96
Population: mITT population consisted of all participants in the ITT population who received at least one dose of study medication and had at least one baseline and post baseline efficacy assessment. As per protocol, data was summarized for the mITT Population using pooled data from participants in this study and TG1101-RMS301 [NCT03277261].
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 543 | 546
weeks | NA [NA to NA] — Median and Inter Quartile Range were not reached due to the low number of participants with events. | NA [NA to NA] — Median and Inter Quartile Range were not reached due to the low number of participants with events.

5. Secondary Outcome: Percentage of Participants With No Evidence of Disease Activity (NEDA)
Description: A participant with NEDA is defined as a participant without relapses confirmed by the IRAP, without MRI activities (no T1 Gd+ lesions and no new/enlarging T2 lesions), and no 12-week CDP. Any evidence of disease activity from Week 24 to Week 96 was counted as not reaching NEDA. Any evidence of disease activity before Week 24 was not counted.
Time Frame: From Week 24 to Week 96
Population: mITT population consisted of all participants in the ITT population who received at least one dose of study medication and had at least one baseline and post baseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 272 | 272
percentage of participants | 43.0 | 11.4
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p < .0001, Regression, Logistic — Logistic regression model with treatment, region, baseline EDSS strata and log transformed baseline MRI lesion counts (T1-unenhancing, T2, Gd-enhancing) as covariates; Odds Ratio (Ublituximab / Teriflunomide) = 7.946, 95% CI 2-sided [4.917 to 12.841]

6. Secondary Outcome: Percentage of Participants With Impaired Symbol Digit Modalities Test (SDMT)
Description: The SDMT involves a simple substitution task using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Responses are done verbally. The administration time is approximately 5 minutes. The total SDMT score for each visit ranging from 0-110 is defined as the total number of correct answers reported in the case report form (CRF), where high scores indicate better outcome. Impaired SDMT is defined as a decrease of at least 4 points from baseline at any post-baseline assessment up to the Week 96 visit.
Time Frame: Baseline to Week 96
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 272 | 272
percentage of participants | 29.0 | 31.6
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p = 0.4290, Regression, Logistic — Logistic regression model with treatment, region, baseline EDSS strata and log transformed baseline MRI lesion counts (T1 unenhancing, T2, Gd enhancing) as covariates; Odds Ratio (Ublituximab / Teriflunomide) = 0.862, 95% CI 2-sided [0.596 to 1.246]

7. Secondary Outcome: Percent Change From Baseline in Brain Volume
Time Frame: Baseline to Week 96
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 235 | 224
percent change | -0.194 [-0.225 to -0.164] | -0.176 [-0.207 to -0.146]
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p = 0.3108, Mixed Model Repeated Measures — Mixed model repeated measures (MMRM) model includes treatment, region, baseline EDSS strata, visit, treatment-by-visit interaction, and baseline volume (cube root transformed) as covariates and an unstructured covariance matrix; Least Squares Mean Difference = -0.018, 95% CI 2-sided [-0.053 to 0.017]

8. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious AE is defined as any untoward medical occurrence that: results in death, is immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, and/or causes a congenital anomaly/birth defect. TEAEs are AEs that start or worsen after receiving the study drug.
Time Frame: From the first dose of study drug through the end of the study (up to approximately 116 weeks)
Population: Safety population included all participants who received at least one dose of study drug (ublituximab or teriflunomide, with corresponding placebos).
Measure: Number; unit: percentage of participants
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 272 | 273
percentage of participants
  TEAEs | 92.3 | 93.8
  TESAEs | 10.3 | 7.7

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through the end of the study (up to approximately 116 weeks)
Description: Safety population included all participants who received at least one dose of study drug (ublituximab or teriflunomide, with corresponding placebos).
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
All-Cause Mortality (participants affected / at risk) | 1/272 | 0/273
Serious Adverse Events (participants affected / at risk) | 28/272 | 21/273
Other Adverse Events (participants affected / at risk) | 234/272 | 233/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ublituximab + Oral Placebo (N=272) | Teriflunomide + IV Placebo (N=273)
Bone marrow toxicity (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Astigmatism (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Retinal degeneration (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Decreased activity (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 3 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 2
Appendicitis (Infections and infestations) | 1 | 0
Chronic hepatitis B (Infections and infestations) | 1 | 0
Complicated appendicitis (Infections and infestations) | 1 | 1
Epididymitis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Chronic tonsillitis (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 2
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial stromal sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Ovarian cystectomy (Surgical and medical procedures) | 1 | 0
Pituitary gland operation (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ublituximab + Oral Placebo (N=272) | Teriflunomide + IV Placebo (N=273)
Lymphopenia (Blood and lymphatic system disorders) | 26 | 2
Anaemia (Blood and lymphatic system disorders) | 9 | 15
Sinus tachycardia (Cardiac disorders) | 20 | 5
Nausea (Gastrointestinal disorders) | 29 | 28
Abdominal pain (Gastrointestinal disorders) | 28 | 12
Diarrhoea (Gastrointestinal disorders) | 25 | 32
Constipation (Gastrointestinal disorders) | 16 | 17
Dyspepsia (Gastrointestinal disorders) | 16 | 15
Toothache (Gastrointestinal disorders) | 16 | 15
Abdominal pain upper (Gastrointestinal disorders) | 15 | 9
Pyrexia (General disorders) | 34 | 14
Influenza like illness (General disorders) | 28 | 7
Chills (General disorders) | 25 | 3
Hyperthermia (General disorders) | 18 | 4
Asthenia (General disorders) | 16 | 20
Fatigue (General disorders) | 15 | 11
Nasopharyngitis (Infections and infestations) | 67 | 54
Respiratory tract infection (Infections and infestations) | 30 | 28
Pharyngitis (Infections and infestations) | 24 | 6
Upper respiratory tract infection (Infections and infestations) | 24 | 25
Respiratory tract infection viral (Infections and infestations) | 22 | 23
Cystitis (Infections and infestations) | 17 | 12
Sinusitis (Infections and infestations) | 17 | 13
Oral herpes (Infections and infestations) | 14 | 16
Rhinitis (Infections and infestations) | 9 | 14
Infusion related reaction (Injury, poisoning and procedural complications) | 19 | 2
Lymphocyte count decreased (Investigations) | 15 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 13
Headache (Nervous system disorders) | 103 | 87
Dizziness (Nervous system disorders) | 16 | 12
Insomnia (Psychiatric disorders) | 21 | 8
Anxiety (Psychiatric disorders) | 16 | 12
Dysmenorrhoea (Reproductive system and breast disorders) | 12 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 9
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 14 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 48
Hypertension (Vascular disorders) | 10 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT03277248/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT03277248/SAP_001.pdf